CLINICAL TRIAL: NCT05121545
Title: A Phase 1 Study of Proton Pencil Beam Scanning GRID for Treatment of Bulky Tumors (ProGRID)
Brief Title: Proton Pencil Beam Scanning GRID for Treatment of Bulky Tumors
Acronym: ProGRID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2161; IRB00289810 (Other: JHM IRB)
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma; Melanoma
Keywords: Spatially-fractionated radiotherapy; GRID-therapy; Proton therapy; Sarcoma; Melanoma; Treatment resistant tumors
MeSH Terms: conditions — Sarcoma; Melanoma

STUDY DESIGN:
Intervention Model Description: This is a single arm phase I study design, evaluating the feasibility (primary endpoint), toxicity (secondary endpoint), and degree of response (exploratory endpoint) after proton GRID therapy in patients with bulky tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pro-GRID treatment Arm (Other): Patients enrolled in this study will receive spatially-fractionated radiotherapy or GRID-therapy, which involves delivering a one-time treatment of high dose radiation to small amounts of tumor in a manner that creates alternating regions of high and low dose radiation within the tumor. Patients will receive 2 (lowest dose) to 18 Gy (highest dose) in a single fraction.
  Interventions: Radiation: Pro-GRID

INTERVENTIONS:
Radiation: Pro-GRID — Study participants will receive a single treatment of Pro-GRID therapy. After which, the participants would be able to resume standard therapy (after one week) and receive additional radiotherapy one month after Pro-GRID therapy, if recommended. Participants will be in the study for one year. Follow-up appointments will be scheduled at 1, 3, 6 and 12 months posttreatment, and may include a history and physical exam, labs and/or a CT scan and toxicity assessments.
  Other Names: Multi-beam proton Pencil Beam Scanning (PBS), termed Pro-GRID

SUMMARY:
This is a single arm, phase I study, evaluating the feasibility, toxicity, and degree of tumor response after novel proton pencil beam scanning (PBS GRID) treatment in patients with bulky tumors that are difficult to manage.

DETAILED DESCRIPTION:
The proton group at Sibley Memorial Hospital has developed a new method for multi-beam proton delivery making it possible to arrange and optimize GRID dosimetry and normal tissue sparing compared to other similar techniques.

In this phase I pilot study, patients with bulky tumors will receive this novel method of GRID-therapy also called spatially-fractionated radiotherapy which involves delivering high dose radiation to small amounts of tumor in a manner that creates alternating regions of high and low dose radiation within the tumor and is often aligned in a grid pattern.

In so doing, this study will ascertain the feasibility, safety and tumor response i.e. shrinkage and resectability of this treatment. Ultimately, the goal is to improve local outcomes of patients with bulky tumors and to offer new treatment options for patients with difficult-to-manage bulky tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically or cytologically confirmed invasive cancer
* Bulky tumor > 7 cm, determined clinically and/or radiographically, at the time of evaluation prior to enrollment
* Treated indicated for palliative intent
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Anticipated treatment deemed safe on pre-review by PI
* For patients with prior Radiation Therapy (RT): Dicoms must be available for dose fusion if overlap anticipated with GRID
* Willing and able to provide informed consent
* Discussion with medical oncology or surgical specialty

Exclusion Criteria:

* Age < 18
* ECOG performance status 3-4
* Planned for definitive, curative management
* For patients with prior RT that overlaps with Pro-GRID: Dicoms not available Pregnant women
* Tumor encasing critical structure, as defined by the treating MD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Pro-GRID intervention as assessed by success of intervention delivery for a number of participants | 1.5 years
  To assess the feasibility of successfully creating treatment plans and delivering a novel proton therapy called Pro-GRID. Feasibility will be determined by a successful intervention delivery for 10 of 12 patients with bulky solid tumors.

SECONDARY OUTCOMES:
Rate of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4) | 3 months post-treatment
  To determine the rate of mild acute toxicity, defined as any CTCAE grade 2 or lower toxicity, and severe acute toxicity, defined as any CTCAE grade 3 or higher toxicity.
Change in rate of treatment response of bulky tumors treated and not treated with proton GRID therapy | 1, 6 and 12 months post-treatment
  To determine the change in response rate for bulky tumors treated and not treated with Proton GRID by Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
Change in degree of treatment response of bulky tumors treated and not treated with proton GRID therapy | 1, 6 and 12 months post-treatment
  Change in degree of treatment response would be measured by RECIST criteria (partial response, complete response, stable disease, or progression of disease).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wright, MD, Principal Investigator — Radiation Oncology, SOM
Locations (1):
- Sibley Memorial Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No